CLINICAL TRIAL: NCT00358995
Title: A New Cognitive Behavioral Therapy to Target Distorted Appraisals Characteristic of Primary Obsessions in Obsessive Compulsive Disorder
Brief Title: A Cognitive Behavioral Therapy of Primary Obsessions in Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H02-80132
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Cognitive Behavioral Therapy; Primary Obsessions; Obsessive Compulsive Disorder; Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Compulsive Personality Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Cognitive Behavior Therapy (CBT) may include keeping a diary of significant events and associated feelings, thoughts and behaviors; questioning and testing cognitions, assumptions, evaluations and beliefs that might be unhelpful and unrealistic; gradually facing activities which may have been avoided; and trying out new ways of behaving and reacting and using relaxation and distraction techniques.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- 2 (Active Comparator): Stress Management Therapy (SMT) includes relaxation, interaction, biofeedback, exercises, such as muscle stretching exercises, yoga, meditation, time management techniques, and many more.
  Interventions: Behavioral: Stress Management Therapy (SMT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Participants will be randomly assigned to either immediate treatment or delayed treatment (three month delay). Participants will then be again be randomly assigned to either Cognitive Behavior Therapy (CBT) or Stress Management Therapy (SMT). The delayed participants (wait list control) will be randomly assigned to either of the two active treatment groups in three months time. Both active treatment conditions involve one hours, individual treatment sessions for 12 consecutive weeks by one of the treating psychologists. All participants will also be asked to complete a package of psychometric questionnaires before treatment.
  Arms: 1
Behavioral: Stress Management Therapy (SMT) — Participants will be randomly assigned to either immediate treatment or delayed treatment (three month delay). Participants will then be again be randomly assigned to either Cognitive Behavior Therapy (CBT) or Stress Management Therapy (SMT). The delayed participants (wait list control) will be randomly assigned to either of the two active treatment groups in three months time. Both active treatment conditions involve one hours, individual treatment sessions for 12 consecutive weeks by one of the treating psychologists. All participants will also be asked to complete a package of psychometric questionnaires before treatment.
  Arms: 2

SUMMARY:
A New Cognitive Behavioral Therapy to Target Distorted Appraisals Characteristic of Primary Obsessions in Obsessive Compulsive Disorder

DETAILED DESCRIPTION:
Participants will be phone-screened to determine broad suitability and interest in being in the study, as well as availability. Following telephone screening, participants will meet with a clinician who will administer a semi-structured interview to determine diagnostic status followed by a more specific standard semi-structured interview to measure symptom strength in those participants who meet diagnostic criteria of OCD (primary obsessions). Participants will then be invited to join the study. Participants will be randomly assigned to either immediate treatment or delayed treatment (three month delay). Participants will then be again be randomly assigned to either Cognitive Behavior Therapy (CBT) or Stress Management Therapy (SMT). The delayed participants (wait list control) will be randomly assigned to either of the two active treatment groups in three months time. Both active treatment conditions involve one hours, individual treatment sessions for 12 consecutive weeks by one of the treating psychologists. All participants will also be asked to complete a package of psychometric questionnaires before treatment. Participants assigned to the delayed treatment condition will be asked to complete these questionnaires again before proceeding to treatment once they have completed the three month wait. The participants will be re-evaluated at the end of treatment, at six months after treatment, and at one year after treatment, using the same assessment procedure.

ELIGIBILITY:
Inclusion Criteria:

involves:

1. a primary diagnosis of OCD,
2. an absence of overt compulsions associated with the primary obsessions,
3. functional impairment due to OCD for at least one year,
4. age range 18-65 years,
5. fluency in spoken and written English,
6. a willingness to undergo random assignment to treatment, and to complete the assigned treatment and planned assignments.

Exclusion Criteria:

1. presence of a severe depressive disorder with suicidal intent requiring immediate intervention,
2. evidence of organic mental disorder, active thought disorder, current alcohol or drug dependence, or mental retardation,
3. concurrent psychological treatment for any axis (i) or (ii) disorder, aside from supportive therapy for depression, and
4. commencement or change in psychotropic medication in the three months prior to initial assessment through to post-treatment assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2002-07; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study is to determine if CBT is more effective than SMT in reducing distorted beliefs and OCD symptoms in study participants post treatment, as well as six and twelve months post treatment. | 12 months

SECONDARY OUTCOMES:
The secondary outcome of the study is to determine if change in appraisals of intrusive thoughts will mediate symptom change during and after treatment (i.e. follow-up). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter McLean, MD, Principal Investigator — The University of British Columbia
Locations (1):
- UBC Hospital, The Anxiety Disorders Clinic, Vancouver, British Columbia, Canada